CLINICAL TRIAL: NCT02097706
Title: A Randomised Double-blind Placebo Controlled Investigation of the Efficacy of a Novel Drug as an Adjunct in Patients With Borderline Personality Disorder
Brief Title: A Novel Drug for Borderline Personality Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Professor, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204-14
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2024-11

CONDITIONS: Borderline Personality Disorder
Keywords: Boderline Personality Disorder; Mental Illness; Cognition
MeSH Terms: conditions — Borderline Personality Disorder; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMDA receptor antagonist (Active Comparator): 20mg/daily for 12 weeks (84 days)
  Interventions: Drug: NMDA receptor antagonist (active drug)
- Placebo tablet (Placebo Comparator): 1 capsule/daily for 12 weeks (84 days)
  Interventions: Other: Lactose packed capsule (inert/inactive arm)

INTERVENTIONS:
Drug: NMDA receptor antagonist (active drug)
  Arms: NMDA receptor antagonist
Other: Lactose packed capsule (inert/inactive arm)
  Arms: Placebo tablet

SUMMARY:
Borderline Personality Disorder (BPD) is one of the most prevalent psychiatric disorders with high morbidity and mortality. It affects the lives of millions worldwide and is often highly incapacitating, leading to significant psychosocial dysfunction. Moreover, nearly all patients have experienced suicidal ideation and about 10% actually commit suicide, a rate almost 50 times higher than in the general population. Mostly young women are at greater risk for the disorder and are three times more likely to be diagnosed with BPD than men.

BPD aetiology is complex and could be explained by both biological and environmental factors. Among the environmental factors, sexual or physical abuse, parental divorce, loss or illnesses are identified as the most common ones. These factors can induce dysfunctional behaviours, which might cause emotional dysregulation, high impulsivity and frequent self- injurious behaviour.

However, there are no pharmacologic interventions that are known to be specifically effective to treat BPD. Therapeutic options for this devastating disorder is still far from adequate for treating acute illness episodes, relapses, and recurrences and in restoring premorbid functioning. In addition, some patients are unable to tolerate existing therapies for BPD, which leads to either frequent changes in medications or to non-adherence. Therefore there is an urgent need for the development of more rapidly effective treatments for BPD.

A growing body of evidence suggests that glutamatergic neurotransmission, in particular N-methyl-D-aspartate (NMDA) subtype may play a role in the pathophysiology of multiple psychiatric disorders. This has led to various clinical trials with glutamate modulating drugs. The trial drug is an uncompetitive NMDA receptor antagonist approved for Alzheimer's disease is increasingly being studied in a variety of non-dementia psychiatric disorders. Results from these studies have proved that the trial drug was safe and well tolerated and has the potential for use in the treatment of psychiatric disorders.

To date, there are no published data on the use of trial drug in the treatment for BPD. Therefore, the investigators intend to study the efficacy of this novel drug as an addition to ongoing therapy with atypical antipsychotics in patients with Borderline Personality Disorder. This study will recruit 150 BPD patients. The patients will be randomly allocated to receive either the study medication (20mg/ day) or placebo via oral administration for twelve weeks. To observe the efficacy of the trial treatment, all participants will be assessed at various time intervals for different borderline and cognitive symptoms.

ELIGIBILITY:
Inclusion criteria

Participants will be eligible to proceed in the study if they meet all of the following criteria (as determined in the screening session):

1. Men and women aged between 18-65 years of age
2. A current diagnosis of BPD, or a score ≥ 8 on Diagnostic Interview for Borderline patients, or a score ≥ 15 on Zanarini Rating Scale for Borderline Personality Disorder
3. Proficient in reading and writing English

Exclusion criteria

Potential participants who meet the criteria for any of the following will be excluded from participating in the study:

1. Clinical evidence of acute delirium or severe head injury
2. Epilepsy or other current seizure disorder, history of seizures or convulsions (not including febrile convulsions), or presence of predisposing factors for epilepsy.
3. Clinically significant hepatic or renal impairment, haematological, or cardiovascular disease.
4. Concomitant use of NMDA antagonists (amantadine, ketamine, dextromethorphan), L-dopa, dopamine agonists or anticholinergics.
5. Lifetime diagnosis of schizophrenia, schizoaffective disorder, substance-induced psychotic disorder or bipolar I disorder (DSM-V).
6. Risk of suicide such that inpatient admission is required, as determined by PI (psychiatrist) on the basis of clinical assessment and baseline BPDSI-IV and/or ZAN-BPD suicide subscale scores.
7. Taking more than 4 psychotropic medications.
8. Planned changes to psychotropic medication or psychotherapy regime.
9. Substance abuse or dependence requiring intervention or rehabilitation in last 3 months.
10. Pregnant or breastfeeding; if of child-bearing age, not using appropriate contraceptive precaution.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Zanarini Rating Scale for Borderline Personality Disorder | Weeks 0, 2, 4, 6, 8, 10, 12
  The Zanarini Rating Scale is a nine-item, validated, clinician-based diagnostic interview. It assesses the severity of DSM-IV-based Borderline personality disorder symptoms. This scale also measures meaningful changes in symptoms over time.

SECONDARY OUTCOMES:
Borderline Evaluation of Severity over Time (BEST) | Weeks 0,2,4,6,8,10,12
  The Borderline Evaluation of Severity over Time (BEST) is a 15-item self-report measure that allows patients with borderline personality disorder (BPD) to rate the degree of impairment or interference from each of the nine BPD criteria over the past two weeks. Each time is rated on a 5-point scale, and scores can range from 12 to 72. Subscales include negative thoughts and feelings, positive behaviours and negative behaviours. The BEST is used to assess the severity of and change in borderline symptoms over the course of treatment.
BPDSI | Baseline and Week 12
  Borderline Personality Disorder Severity Index-IV (BPDSI-IV)
Cogstate (cognitive assessment) | Baseline and Week 12
  Cogstate tests have been designed, developed and validated to both identify and measure cognitive impairment, and to track or monitor cognitive change. The tasks use novel visual and verbal stimuli to ensure assessment is culture-neutral and not limited by a participant's level of education.

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni AM, MBBS,MPM,FRANZCP,PhD, Principal Investigator — Bayside Health, Alfred Hospital
Locations (1):
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174
- [Derived] Kulkarni J, Thomas N, Hudaib AR, Gavrilidis E, Grigg J, Tan R, Cheng J, Arnold A, Gurvich C. Effect of the Glutamate NMDA Receptor Antagonist Memantine as Adjunctive Treatment in Borderline Personality Disorder: An Exploratory, Randomised, Double-Blind, Placebo-Controlled Trial. CNS Drugs. 2018 Feb;32(2):179-187. doi: 10.1007/s40263-018-0506-8. PMID 29549516